CLINICAL TRIAL: NCT02959463
Title: Phase I Trial of Adjuvant Pembrolizumab After Radiation Therapy for Lung-Intact Malignant Pleural Mesothelioma
Brief Title: Pembrolizumab After Radiation Therapy in Treating Patients With Pleural Malignant Mesothelioma
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2015-0856; NCI-2016-01923 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2015-0856 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2016-11-07; First posted 2016-11-09 (Estimated); Results first posted 2025-11-13 (Actual); Last update posted 2025-11-13 (Actual); Status verified 2025-10

CONDITIONS: Pleural Malignant Mesothelioma
MeSH Terms: conditions — Mesothelioma, Malignant | interventions — pembrolizumab; Radiotherapy; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 1 (hemithoracic radiation therapy, pembrolizumab) (Experimental): Patients undergo hemithoracic radiation therapy. After radiation therapy, patients receive pembrolizumab IV over about 30 minutes on day 1. Courses repeat every 3 weeks for up to 2 years in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Laboratory Biomarker Analysis; Biological: Pembrolizumab; Radiation: Radiation Therapy
- Cohort 2 (palliative radiation therapy, pembrolizumab) (Experimental): Patients undergo palliative radiation therapy over 1-3 weeks to only the region of palliation (a region that does not include the entire side of the chest or thorax). After radiation therapy, patients receive pembrolizumab IV over about 30 minutes on day 1. Courses repeat every 3 weeks for up to 2 years in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Laboratory Biomarker Analysis; Radiation: Palliative Radiation Therapy; Biological: Pembrolizumab

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Radiation: Palliative Radiation Therapy — Undergo palliative radiation therapy
  Arms: Cohort 2 (palliative radiation therapy, pembrolizumab)
Biological: Pembrolizumab — Given IV
  Other Names: Keytruda; Lambrolizumab; MK-3475; SCH 900475
Radiation: Radiation Therapy — Undergo hemithoracic radiation therapy
  Other Names: Cancer Radiotherapy; Irradiate; Irradiated; irradiation; Radiation; Radiotherapeutics; RADIOTHERAPY; RT; Therapy, Radiation
  Arms: Cohort 1 (hemithoracic radiation therapy, pembrolizumab)

SUMMARY:
This phase I trial studies the side effects and best way to give pembrolizumab after radiation therapy in treating patients with pleural malignant mesothelioma. Radiation therapy uses high energy radiation to kill tumor cells and shrink tumors. Immunotherapy with monoclonal antibodies, such as pembrolizumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Giving pembrolizumab after radiation therapy may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the safety and tolerability of pembrolizumab administered after radiation therapy in patients with malignant pleural mesothelioma (MPM) who have not undergone extrapleural pneumonectomy.

SECONDARY OBJECTIVES:

I. To assess progression-free and overall survival (progression free survival [PFS] and overall survival [OS], respectively) in patients receiving pembrolizumab after radiation therapy for malignant pleural mesothelioma (MPM).

EXPLORATORY OBJECTIVES:

I. To evaluate biomarkers of interest, including cytokines, measurements of T-cell activation, and serum exosome micro ribonucleic acid (RNA)s with the delivery of pembrolizumab after radiation therapy for MPM.

OUTLINE: Patients are assigned to 1 of 2 cohorts.

COHORT 1: Patients undergo hemithoracic radiation therapy.

COHORT 2: Patients undergo palliative radiation therapy over 1-3 weeks to only the region of palliation (a region that does not include the entire side of the chest or thorax).

After radiation therapy, both cohorts receive pembrolizumab intravenously (IV) over about 30 minutes on day 1. Courses repeat every 3 weeks for up to 2 years in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days, every 6 weeks for 48 weeks, then every 12 weeks for up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a histologic diagnosis of malignant pleural mesothelioma, with histologic diagnosis from the pleura or relevant lymph node stations, including mediastinal, hilar, or supraclavicular lymph nodes
* Be willing and able to provide written informed consent/assent for the trial
* Have measurable or non-measurable disease per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1; however, note that patients in Cohort 1 that have undergone an R0 resection will be eligible for the trial
* Have a performance status of 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) performance scale
* Absolute neutrophil count (ANC) >=1,500 /mcL (within 10-15 days of treatment initiation)
* Platelets >= 100,000 /mcL (within 10-15 days of treatment initiation)
* Hemoglobin >= 9 g/dL or >= 5.6 mmol/L without transfusion or erythropoietin (EPO) dependency (within 7 days of assessment) (within 10-15 days of treatment initiation)
* Serum creatinine =< 1.5 X upper limit of normal (ULN) or measured or calculated creatinine clearance (glomerular filtration rate [GFR] can also be used in place of creatinine or creatinine clearance [CrCl]) >= 60 mL/min for subject with creatinine levels > 1.5 X institutional ULN (within 10-15 days of treatment initiation)
* Serum total bilirubin =< 1.5 X ULN or direct bilirubin =< ULN for subjects with total bilirubin levels > 1.5 ULN (within 10-15 days of treatment initiation)
* Aspartate aminotransferase (AST) serum glutamic oxaloacetic transaminase (SGOT) and alanine aminotransferase (ALT) serum glutamic pyruvic transaminase (SGPT) =< 2.5 X ULN or =< 5 X ULN for subjects with liver metastases (within 10-15 days of treatment initiation)
* Albumin >= 2.5 mg/dL (within 10-15 days of treatment initiation)
* International normalized ratio (INR) or prothrombin time (PT) =< 1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or partial thromboplastin time (PTT) is within therapeutic range of intended use of anticoagulants (within 10-15 days of treatment initiation)
* Activated partial thromboplastin time (aPTT) =< 1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants (within 10-15 days of treatment initiation)
* Female subject of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication; if the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
* Female subjects of childbearing potential should be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 120 days after the last dose of study medication; subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year
* Male subjects should agree to use an adequate method of contraception starting with the first dose of study therapy through 120 days after the last dose of study therapy
* COHORT 1 (PATIENTS RECEIVING HEMITHORACIC RADIATION THERAPY)
* Patients must not have evidence of metastatic disease per positron emission tomography (PET)/ computed tomography (CT) scan; mediastinal lymph node involvement is acceptable
* Patients will have received at least 2 cycles of induction chemotherapy with pemetrexed/cisplatin or pemetrexed/carboplatin
* Forced expiratory volume in 1 second (FEV1) >= 30% of predicted postoperative (ppoFEV1, as if patient underwent a pneumonectomy)
* Diffusing capacity of the lungs for carbon monoxide (DLCO) > 35% predicted
* Patients must be assessed to be a suitable candidate for hemithoracic radiation therapy per the treating radiation oncologist; if the patient undergoes pleurectomy/decortication, they must initiate hemithoracic radiation therapy within 4 months of the surgery date; patients that do not meet the dose constraints outlined below will be removed from the study prior to radiation therapy
* COHORT 2 INCLUSION CRITERIA
* Patients must be assessed to be a suitable candidate for radiation therapy by the treating radiation oncologist; patients that do not meet the dose constraints outlined below will be removed from the study prior to radiation therapy
* Any prior number of prior therapies, including prior immunotherapy, is allowed
* Patient must have prior treatment with a platinum plus pemetrexed regimen

Exclusion Criteria:

* Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of treatment
* Has a diagnosis of immunodeficiency; note that patients should not receive steroids during pembrolizumab administration
* Has a known history of active tuberculosis (TB) (Bacillus tuberculosis)
* Hypersensitivity to pembrolizumab or any of its excipients
* Has had a prior anti-cancer monoclonal antibody (mAb) within 4 weeks prior to study day 1 or who has not recovered (i.e., =< grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier
* Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study day 1 and who have not recovered adequately from this treatment (=< grade 2 toxicity at the time of enrollment)
* Has a known additional malignancy that is progressing or requires active treatment; patients with a stage I-III cancer that has been cured over two years ago are not excluded in the study
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis; subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment; this exception does not include carcinomatous meningitis which is excluded regardless of clinical stability
* Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs); replacement therapy (e.g. thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment
* Has a history of (non-infectious) pneumonitis that required steroids or current pneumonitis
* Has an active infection requiring systemic therapy
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment
* Has a known history of human immunodeficiency virus (HIV) (HIV 1/2 antibodies)
* Has known active hepatitis B (e.g., hepatitis B surface antigen [HBsAg] reactive) or hepatitis C (e.g., hepatitis C virus [HCV] ribonucleic acid [RNA] [qualitative] is detected)
* Has received a live vaccine within 30 days of planned start of study therapy

  * Note: seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist) are live attenuated vaccines, and are not allowed
* Evidence of interstitial lung disease
* COHORT 1 EXCLUSION CRITERIA
* Patients undergoing an extrapleural pneumonectomy (EPP); lung sparing surgeries, such as pleurectomy/decortication, are acceptable
* Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent
* COHORT 2 EXCLUSION CRITERIA
* Patients in which hemithoracic radiation therapy is planned
* Patients who have received EPP for mesothelioma
* COHORTS 1 AND 2 EXCLUSION CRITERIA
* Patients with inherited syndromes associated with hypersensitivity to ionizing radiation, specifically patients with known history of ataxia-telengiectasia, Nijmegen breakage syndrome

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2024-11-15 (Actual); Study Completion 2025-12-31 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Ning, MD, MPH, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Single center trial that recruited patients at one hospital site (MD Anderson Cancer Center, Houston, TX)
Groups:
- Cohort 1: Patient with lung intact to receive hemithoracic radiation therapy for definitive intent
- Cohort 2: Patients with lung intact to receive non-hemithoracic radiation therapy(palliative radiation therapy)
Period: Overall Study
Arm/Group | Cohort 1 | Cohort 2
Started | 12 | 12
Completed | 9 | 11
Not Completed | 3 | 1
Not completed — Adverse Event | 1 | 1
Not completed — Death | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 4 | 8
  >=65 years | 8 | 8 | 16
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 5 | 8
  Male | 9 | 7 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 2
  Not Hispanic or Latino | 12 | 10 | 22
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 11 | 10 | 21
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 2 | 2
Region of Enrollment [Number; unit: participants]
  United States | 12 | 12 | 24

OUTCOME MEASURES:

1. Primary Outcome: Safety/Toxicity
Description: To determine the safety and tolerability of pembrolizumab administered after radiation therapy in patients with MPM. The primary endpoint was "unaccepable" high grade adverse events (AEs) from baseline to 4-month after the start of radiation therapy.
Time Frame: Baseline to 4-months after the start of radiation therapy
Measure: Number; unit: participants
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 12 | 12
participants | 0 | 0

2. Secondary Outcome: Overall Survival (OS)
Description: To assess overall survival (OS) in patients receiving Pembrolizumab after radiation therapy for MPM.
Time Frame: Every 6 weeks (42 +/- 7 days) until to 48 weeks, then every 12 weeks (+/- 7 days) to 5 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 12 | 12
months | 12.2 [7.7 to 23.6] | 16.3 [6.3 to 22.2]

3. Secondary Outcome: Progression-Free Survival (PFS)
Description: To assess progression-free survial (PFS) in patients receiving Pembrolizumab after radiation therapy for MPM.
Time Frame: Every 6 weeks (42 +/- 7 days) until to 48 weeks, then every 12 weeks (+/- 7 days) to 5 years
Measure: Mean (95% Confidence Interval); unit: months
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 12 | 12
months | 7.7 [4.2 to 19.8] | 4 [3.3 to 11.4]

ADVERSE EVENTS:
Time Frame: Baseline to 4-months after radiation therapy up to 5 years
Description: Adverse events (AEs) and serious adverse events (SAEs) are monitered from the baseline to 4-months after Radiation therapy
Arm/Group | Cohort 1 | Cohort 2
All-Cause Mortality (participants affected / at risk) | 11/12 | 12/12
Serious Adverse Events (participants affected / at risk) | 6/12 | 3/12
Other Adverse Events (participants affected / at risk) | 12/12 | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (N=12) | Cohort 2 (N=12)
Death NOS (General disorders) | 1 (1) | 0 (0)
Dysphagia (General disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Esophagitis (General disorders) | 1 (1) | 0 (0)
Gastritis (General disorders) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 5 (5) | 0 (0)
Infections and infestations - Other (Infections and infestations) | 1 (2) | 0 (0)
Creatinine increased (Investigations) | 0 (0) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Acute Kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0)
Tracheal mucositis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Thromboembolic event (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (N=12) | Cohort 2 (N=12)
Anemia (Blood and lymphatic system disorders) | 6 (12) | 8 (8)
Blood and lymphatic system disorders-Other, specify (Blood and lymphatic system disorders) | 3 (8) | 5 (8)
Edema Limbs (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Atrial Flutter (Cardiac disorders) | 0 (0) | 1 (1)
Heart failure (Cardiac disorders) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 1 (3) | 0 (0)
Ear Pain (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Endocrine disorders-Other, (Endocrine disorders) | 1 (1) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 1 (1)
Hypothyroidism (Endocrine disorders) | 1 (5) | 2 (2)
Blurred vision (Eye disorders) | 0 (0) | 1 (1)
Eyelid function disorder (Eye disorders) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (2) | 0 (0)
Alanine aminotransferase increased (Gastrointestinal disorders) | 2 (2) | 0 (0)
Aspartate aminotransferase increased (Gastrointestinal disorders) | 3 (3) | 1 (1)
Constipation (Gastrointestinal disorders) | 4 (5) | 3 (3)
Diarrhea (Gastrointestinal disorders) | 1 (2) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 8 (11) | 5 (6)
Esophagitis (Gastrointestinal disorders) | 6 (7) | 4 (5)
Nausea (Gastrointestinal disorders) | 4 (8) | 4 (5)
Vomiting (Gastrointestinal disorders) | 4 (9) | 1 (1)
Chills (General disorders) | 1 (1) | 0 (0)
Edema Limbs (General disorders) | 1 (1) | 1 (1)
Fatigue (General disorders) | 11 (25) | 9 (16)
Fever (General disorders) | 1 (1) | 0 (0)
Gait disturbance (General disorders) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 2 (2) | 2 (2)
Localized edema (General disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 8 (17) | 4 (5)
Papulopustular rash (Infections and infestations) | 1 (1) | 0 (0)
Infections and infestations-Other,specify (Infections and infestations) | 1 (2) | 0 (0)
Lung infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Dermatitis radiation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 1 (1) | 1 (2)
Alkaline phosphatase increased (Investigations) | 2 (4) | 2 (3)
Alanine aminotansferase increased (Investigations) | 2 (2) | 0 (0)
Aspartate aminotansferase increased (Investigations) | 3 (3) | 1 (1)
Creatinine increased (Investigations) | 4 (5) | 4 (4)
Lymphocyte count decreased (Investigations) | 3 (14) | 1 (1)
Neutrophil count decreased (Investigations) | 0 (0) | 1 (1)
Weight loss (Investigations) | 2 (2) | 4 (4)
White blood cell decreased (Investigations) | 1 (1) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 6 (9) | 3 (3)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 3 (3) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypermagnesemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperuricemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (2) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (3) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Cognitive disturbance (Nervous system disorders) | 1 (1) | 0 (0)
Concentration impairment (Nervous system disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 2 (2) | 1 (1)
Dysgeusia (Nervous system disorders) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 1 (1) | 1 (1)
Nervous system disorders-Other, specify (Nervous system disorders) | 0 (0) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 2 (2) | 0 (0)
Paresthesia (Nervous system disorders) | 2 (2) | 1 (1)
Presyncope (Nervous system disorders) | 2 (2) | 0 (0)
Stroke (Nervous system disorders) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 3 (3) | 0 (0)
Depression (Psychiatric disorders) | 3 (3) | 1 (1)
Insomnia (Psychiatric disorders) | 2 (2) | 0 (0)
Acute Kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 10 (15) | 11 (12)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 10 (16) | 8 (11)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (3)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Breast Pain (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Rash acneiform (Skin and subcutaneous tissue disorders) | 3 (4) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin and subcutaneous tissue disorders- Other,specify (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Social circumstances-Other, specify (Social circumstances) | 1 (2) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-06-07): https://cdn.clinicaltrials.gov/large-docs/63/NCT02959463/Prot_SAP_000.pdf